CLINICAL TRIAL: NCT02478346
Title: Yellow 560 Microscope for Intraoperative Visualization of Fluorescein Stained Intracranial Lesions
Acronym: Fluoescein
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 684812
Record Dates: First submitted 2015-05-27; First posted 2015-06-23 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Cerebrovascular Disorders; Intracranial Neoplasms
MeSH Terms: conditions — Cerebrovascular Disorders; Brain Neoplasms | interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Experimental): All patients enrolled in the study will prepare for surgery as per standard neurosurgical indications, procedures and institution protocols. At the time of the anesthesia induction, with the patient under general anesthesia, Fluorescein Sodium 10% (100mg/1mL) at a dose of 500mg (100mg/ml) will be administered intravenously (the optimal dosage will be determined within the study as the most minimal dose for adequate visualization will be used).
  Interventions: Drug: Fluorescein Sodium

INTERVENTIONS:
Drug: Fluorescein Sodium — Conventional microsurgical and biopsy procedures and techniques including histopathology and intraoperative imaging will be performed through the completion of the surgery. The surgeon will resect and remove what he believes is the tumor based on previously known criteria (standards of care) regardless of what the Fluorescein angiography demonstrates. For vascular lesions, fluorescein sodium 10% (100mg/1mL) will be injected and used to assess its application after the conventional methods have confirmed the exclusion of the aneurysm. No patient's care will be affected by the results of the Fluorescein angiography.

SUMMARY:
This study focuses on implementing Yellow 560 for the direct intraoperative visualization of Fluorescein Sodium stained intracranial lesions to facilitate extend of surgery, develop better treatment protocols, and improve the prognosis of a wide array of neurosurgical diseases. More specifically, for the patients who are undergoing surgical intervention for the treatment of their brain aneurysm, tumor, arteriovenous malformation or fistula, the investigators will inject the dye intraoperatively to assess for residual aneurysm, tumor or in general residual lesion which must be corrected.

DETAILED DESCRIPTION:
The research design is a prospective clinical study. All patients enrolled in the study will prepare for surgery as per standard neurosurgical indications, procedures and institution protocols. At the time of the anesthesia induction, with the patient under general anesthesia, Fluorescein Sodium 10% (100mg/1mL) at a dose of 500mg (100mg/ml) will be administered intravenously (the optimal dosage will be determined within the study as the most minimal dose for adequate visualization will be used). Surgery will continue with the aid of the Yellow 560 microscope with a minimum delay of 10 minutes after injection to reduce the amount of leakage of Fluorescein Sodium into the surrounding tissue.

Conventional microsurgical and biopsy procedures and techniques including histopathology and intraoperative imaging will be performed through the completion of the surgery. The surgeon will resect and remove what he believes is the tumor based on previously known criteria (standards of care) regardless of what the Fluorescein angiography demonstrates. For vascular lesions, fluorescein sodium 10% (100mg/1mL) will be injected and used to assess its application after the conventional methods have confirmed the exclusion of the aneurysm. No patient's care will be affected by the results of the Fluorescein angiography.

No other additional neurosurgical instruments will be used. Patients will be treated post-operatively with conventional adjunctive therapies and imaging as deemed necessary by the attending neurosurgeon for the evaluation of extent of surgery. Follow-up data (including post-operative images assessing outcomes and complications) will be collected on all patients on standard post-operative visits. Intra-operative films or recordings and all patient data may be saved and used according to HIPAA allowances.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18)
* Diagnosed by preoperative imaging modalities to have a brain tumor (including metastatic brain tumors) or vascular lesions (aneurysm, arteriovenous malformation or arteriovenous fistula) requiring surgical intervention.
* The patient is determined by a board certified neurosurgeon to have a tumor or vascular lesion that would take up fluorescein
* Patient or legally authorized representative provides written informed consent to enroll in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intracerebral lesion | Particpants will be followed from enrollment into study which include atleast to 2 images and any other image done up to 1 year of scheudled follow up.
  The main outcome measure of the study would be a comparison between patient pre-operative and post-operative images to evaluate the potential utility of using Fluorescein Sodium and the Yellow 560 microscope to aid in the treatment of intracranial tumors and vascular lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Gandhi, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

REFERENCES:
- [Background] 1. Ciardella AP, Kaufman SR, Yannuzzi LA. The use of fluorescein angiography in acquired macular diseases. In: Tasman W, Jaeger EA, eds. Foundations of Clinical Ophthalmology. 15th ed. Philadelphia, Pa: Lippincott Williams & Wilkins; 2009:chap 113F.
- [Background] 2. Dithmar, Stefan, Holz, Frank G. Fluorescence Angiography in Ophthalmology. 2008, X, 224 p. 541 illus. in color.
- [Background] 3. Maguire JI, Federman JL. Intravenous fluorescein angiography. In: Tasman W, Jaeger EA, eds. Duane's Ophthalmology. 15th ed. Philadelphia, Pa: Lippincott Williams & Wilkins; 2009:chap 44.